CLINICAL TRIAL: NCT03530215
Title: Evaluation of Reporting of Cardio-vascular Adverse Events With Antineoplastic and Immunomodulating Agents (EROCA)
Acronym: EROCA
Status: Completed | Type: Observational
Sponsor: Groupe Hospitalier Pitie-Salpetriere (Other)
Responsible Party: Principal Investigator, Joe Elie Salem, Assistant director, clinical investigation center Paris Est, Groupe Hospitalier Pitie-Salpetriere
Other Study IDs: CIC1421-18-12
Record Dates: First submitted 2018-05-08; First posted 2018-05-21 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: Cardiac Disease; Cancer
Keywords: Cardiotoxicity; Antineoplastic and immunomodulating agents
MeSH Terms: conditions — Heart Diseases; Neoplasms; Cardiotoxicity | interventions — Antineoplastic Agents; Immunomodulating Agents

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Adverse Events with Antineoplastic and immunomodulating agents: Cases reported in the World Health Organization (WHO) and the French pharmacovigilance database of patients treated by Antineoplastic and immunomodulating agents, with a chronology compatible with the drug toxicity
  Interventions: Drug: Antineoplastic and Immunomodulating Agents

INTERVENTIONS:
Drug: Antineoplastic and Immunomodulating Agents — Antineoplastic agents, endocrine therapy, immunostimulants and immunosuppressants drugs included in the ATC classification L

SUMMARY:
Antineoplastic and immunomodulating agents may lead to various cardio-vascular adverse reactions. This study investigates reports of cardio-vascular toxicities for treatment including Anatomical Therapeutic Chemical (ATC) classification L (antineoplastic agents, endocrine therapy, immunostimulants, and immunosuppressants drugs) in the World Health Organization's (WHO) global database of individual safety case reports (VigiBase).

DETAILED DESCRIPTION:
Antineoplastic therapies are responsible of a wide range of cardio-vascular side effects.The investigators use VigiBase, the World Health Organization (WHO) database of individual safety case reports, to identify cases of cardiovascular adverse drug reactions following treatment with antineoplastic and immunomodulating agents

ELIGIBILITY:
Inclusion Criteria:

* Case reported in the World Health Organization (WHO) database of individual safety case reports to 30/04/2018
* Adverse events reported were including the MedDRA terms: Cardiac and vascular investigations (excl enzyme tests) (HLGT), Vascular disorders (SOC), Skeletal and cardiac muscle analyses (HLT), Sudden death (PT), Sudden cardiac death (PT), Cardiac disorders (SOC), Cardiac arrhythmias (HLGT), Cardiac disorder signs and symptoms (HLGT), Cardiac neoplasms (HLGT), Cardiac valve disorders (HLGT), Congenital cardiac disorders (HLGT), Coronary artery disorders (HLGT), Endocardial disorders (HLGT), Heart failures (HLGT), Myocardial disorders (HLGT), Pericardial disorders (HLGT)
* Patients treated with Antineoplastic and immunomodulating agents included in the ATC L.

Exclusion Criteria:

* Chronology not compatible between the drug and the toxicity

Ages: 0 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients treated with Antineoplastic and immunomodulating agents
Sampling Method: Non-Probability Sample
Enrollment: 500000 (Actual)
Dates: Start 2018-05-02 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2023-04-08 (Actual)

PRIMARY OUTCOMES:
Cardio-vascular toxicity of antineoplastic and immunomodulating agents | Case reported in the World Health Organization (WHO) of individual safety case reports to September 2018
  Identification and report of cardio-vascular toxicities of antineoplastic and immunomodulating agents. The research includes the report with MedDRA terms: SOC Cardiac Disorders, SOC Vascular Disorders, Sudden death (PT), Cardiac and vascular investigations (excl enzyme tests) (HLGT), Skeletal and cardiac muscle analyses (HLT)

SECONDARY OUTCOMES:
Causality assessment of reported cardiovascular events according to the WHO system | Case reported in the World Health Organization (WHO) of individual safety case reports to September 2018
Description of the type of cardiotoxicity depending on the category of antineoplastic and immunomodulating agents | Case reported in the World Health Organization (WHO) of individual safety case reports to September 2018
Description of the duration of treatment when the toxicity happens | Case reported in the World Health Organization (WHO) of individual safety case reports to September 2018
Description of the drug-drug interactions associated with adverse events | Case reported in the World Health Organization (WHO) of individual safety case reports to September 2018
Description of the pathologies (cancer) for which the incriminated drugs have been prescribed | Case reported in the World Health Organization (WHO) of individual safety case reports to September 2018
Description of the population of patients having a cardio-vascular adverse event | Case reported in the World Health Organization (WHO) of individual safety case reports to September 2018

CONTACTS AND LOCATIONS:
Locations (1):
- AP-HP, Pitié-Salpêtrière Hospital,Department of Pharmacology, CIC-1421, Pharmacovigilance Unit, INSERM., Paris, France

REFERENCES:
- [Derived] Salem JE, Nguyen LS, Moslehi JJ, Ederhy S, Lebrun-Vignes B, Roden DM, Funck-Brentano C, Gougis P. Anticancer drug-induced life-threatening ventricular arrhythmias: a World Health Organization pharmacovigilance study. Eur Heart J. 2021 Oct 7;42(38):3915-3928. doi: 10.1093/eurheartj/ehab362. PMID 34370839
- [Derived] Xiao L, Salem JE, Clauss S, Hanley A, Bapat A, Hulsmans M, Iwamoto Y, Wojtkiewicz G, Cetinbas M, Schloss MJ, Tedeschi J, Lebrun-Vignes B, Lundby A, Sadreyev RI, Moslehi J, Nahrendorf M, Ellinor PT, Milan DJ. Ibrutinib-Mediated Atrial Fibrillation Attributable to Inhibition of C-Terminal Src Kinase. Circulation. 2020 Dec 22;142(25):2443-2455. doi: 10.1161/CIRCULATIONAHA.120.049210. Epub 2020 Oct 23. PMID 33092403
- [Derived] Salem JE, Ederhy S, Lebrun-Vignes B, Moslehi JJ. Cardiac Events Associated With Chimeric Antigen Receptor T-Cells (CAR-T): A VigiBase Perspective. J Am Coll Cardiol. 2020 May 19;75(19):2521-2523. doi: 10.1016/j.jacc.2020.02.070. No abstract available. PMID 32408984
- [Derived] Alexandre J, Salem JE, Moslehi J, Sassier M, Ropert C, Cautela J, Thuny F, Ederhy S, Cohen A, Damaj G, Vilque JP, Plane AF, Legallois D, Champ-Rigot L, Milliez P, Funck-Brentano C, Dolladille C. Identification of anticancer drugs associated with atrial fibrillation: analysis of the WHO pharmacovigilance database. Eur Heart J Cardiovasc Pharmacother. 2021 Jul 23;7(4):312-320. doi: 10.1093/ehjcvp/pvaa037. PMID 32353110
- [Derived] Salem JE, Manouchehri A, Bretagne M, Lebrun-Vignes B, Groarke JD, Johnson DB, Yang T, Reddy NM, Funck-Brentano C, Brown JR, Roden DM, Moslehi JJ. Cardiovascular Toxicities Associated With Ibrutinib. J Am Coll Cardiol. 2019 Oct 1;74(13):1667-1678. doi: 10.1016/j.jacc.2019.07.056. PMID 31558250